CLINICAL TRIAL: NCT00193986
Title: Assessment of Prepulse Inhibition for Shock Pain Reduction- Ventricular
Brief Title: Assessment of Prepulse Inhibition for Shock Pain Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Dr. Douglas Cameron (Unknown); Abbott Medical Devices (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 04-0252-B
Record Dates: First submitted 2005-09-08; First posted 2005-09-19 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-09

CONDITIONS: Pain Awareness From ICD Shocks
Keywords: Prepulse; Defibrillator

INTERVENTIONS:
Device: Arbitrary Waveform Defibrillator

SUMMARY:
Patient tolerance of pain from discharges of implantable cardioverter defibrillators (ICD's) is highly variable. It can be influenced by psychological factors, physical condition and the number of shocks delivered.

It has been shown that cutaneous pain perception can be reduced by delivery of a weak , low voltage pulse (prepulse)prior to the delivery of a stronger shock.

A prepulse delivered before a high voltage ICD shock will decrease discomfort compared to a shock of equal energy without a prepulse.

ELIGIBILITY:
Inclusion Criteria:

18+ Approved indication for implantation of an ICD Able and willing to provide informed consent Independently complete and understand the Mini Mental State Evaluation

Exclusion Criteria:

Pregnancy Cannot understand English or French Contraindicated for defibrillation testing because of risk of thromboembolism Deaf or hard of hearing, making the acute testing difficult to conduct having pain or anxiety to the extent that, in the opinion of the investigator, the results would be confounded.

Having a Class I bradycardia pacing indication, requiring ongoing pacing support.

Visual problems which preclude reading the computer screen for the VAS test Severe musculoskeletal disorder that makes it difficult to undergo testing in the recumbent position Do not achieve a score >24/30 on a Mini Mental State Exam

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Assessment from pain perception from a shock preceded by a prepulse compared to a non prepulsed shock

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Cameron, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada